CLINICAL TRIAL: NCT00554320
Title: Effect of Repetitive Transcranial Direct Current Stimulation (tDCS) on Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Bradford W. Fenton, MD, PhD; Director, Summa Helath System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP07066
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Pelvic Pain; Interstitial Cystitis; Post Traumatic Stress Disorder; Fibromyalgia; Irritable Bowel Syndrome
Keywords: vulvodynia; painful bladder syndrome; myofascial pain syndrome; pelvic floor tension myalgia
MeSH Terms: conditions — Cystitis, Interstitial; Stress Disorders, Post-Traumatic; Fibromyalgia; Irritable Bowel Syndrome; Vulvodynia; Myofascial Pain Syndromes | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): During each session, the anode electrode will be placed on the motor cortex (contralateral to the most [or predominant] painful side [or the side where the symptoms begin or the left as a default]) and the cathode will be placed over the contralateral supraorbital area. In active tDCS subjects, 1 mA of transcranial direct current stimulation will be applied for 30 minutes.
  Interventions: Procedure: tDCS
- C (Placebo Comparator): For sham-controlled tDCS subjects, the same montage will be used; however current will be applied only for 30 seconds.
  Interventions: Procedure: tDCS

INTERVENTIONS:
Procedure: tDCS — During each session, the anode electrode will be placed on the motor cortex (contralateral to the most [or predominant] painful side [or the side where the symptoms begin or the left as a default]) and the cathode will be placed over the contralateral supraorbital area. In active tDCS subjects, 1 mA of transcranial direct current stimulation will be applied for 30 minutes.
  Arms: A
Procedure: tDCS — For sham-controlled tDCS subjects, the same montage will be used; however current will be applied only for 30 seconds.
  Arms: C

SUMMARY:
We will rigorously test whether modulation of the motor cortex by transcranial direct current stimulation (tDCS) is an effective treatment for patients with chronic pelvic pain through the following specific aims:

A) The primary aim of this study is to determine whether transcranial direct current stimulation applied to the motor cortex in patients with chronic pelvic pain induces a significant decrease in the pain or symptoms as compared with sham tDCS. We will also measure changes in the clinical symptom scores of multiple pelvic organs, drug intake (narcotic), anxiety, depression, traumatic stress, as well as overall improvement in the quality of life to assess the effects of this treatment.

B) Determine the duration of the clinical effects of tDCS. We will therefore compare the amelioration of pain and related symptoms between active and sham tDCS for one year following treatment.

C) Determine whether tDCS changes the threshold for pain detection as compared with sham tDCS. Patients with chronic pelvic pain have a lower threshold for pain as compared to healthy subjects and we hypothesized that this threshold will increase after stimulation with tDCS.

D) Finally, we will examine whether 5 days of tDCS treatment is safe for use in chronic pelvic pain patients. Safety will be assessed through neuropsychological tests and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be females between 18 and 55 years of age.
* Subjects must have a current VAS for pelvic pain of 5 or more.

Exclusion Criteria:

* Known pelvic malignancy.
* Patients with major depression with suicidal risk as clinically defined.
* Patients with other known, uncontrolled neuropsychiatric disorders.
* Abnormal neurological examination other than as signs of the condition studied in the present protocol.
* Contraindication to tDCS:
* A history of unmanaged substance abuse or dependence within the last 6 months.
* A history of previous treatment with tDCS.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Patient Global Assessment (PGA): | 2 weeks
Visual analog scale (VAS) for pain: | 2 weeks

SECONDARY OUTCOMES:
Interstitial cystitis symptom index: | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bradford W Fenton, MD, PhD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States